CLINICAL TRIAL: NCT04557345
Title: Evaluation of the Inflammatory Response and Long-term Calcification in Post-operated Aortic Valve Replacement Patients.
Brief Title: Evaluation of the Inflammatory Response in Post-operated Aortic Valve Replacement Patients.
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Maria Elena Soto, MsC and PhD, Principal Investigator, Instituto Nacional de Cardiologia Ignacio Chavez
Other Study IDs: 17-1033
Record Dates: First submitted 2020-08-28; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Aortic Valve Disease; Aortic Valve Stenosis; Aortic Valve Calcification; Prosthetic Valve Malfunction
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis; Aortic Valve, Calcification of

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Biological prostheses INC: Prosthetic valve manufactured in the National Institute of Cardiology "Ignacio Chávez".
  Interventions: Diagnostic Test: Determination of cytokines; Diagnostic Test: Two-dimensional transthoracic echocardiogram
- Imported Biological aortic prostheses: St Jude EPIC and Carpentier-Edwards Perimount
  Interventions: Diagnostic Test: Determination of cytokines; Diagnostic Test: Two-dimensional transthoracic echocardiogram
- Mechanical prostheses: St Jude Masters HP, Carbomedics Standart, ON-X Life Technologies, Edwards Mira, Carbomedics Orbis, Medtronic Hall and Medtronic ATS.
  Interventions: Diagnostic Test: Determination of cytokines; Diagnostic Test: Two-dimensional transthoracic echocardiogram
- Control: In subjects who come to donate blood products altruistically, in the blood bank service of the INC, with prior informed consent, the subjects will be matched with PO patients of CVA by age and gender.
  Interventions: Diagnostic Test: Determination of cytokines; Diagnostic Test: Two-dimensional transthoracic echocardiogram

INTERVENTIONS:
Diagnostic Test: Determination of cytokines — Subsequently, a blood sample will be taken from which the processing will be as follows: 6 ml of peripheral blood will be taken in tubes with a yellow cap and inert gel and clot retractor, immediately afterward it will be placed on ice, it will be transported to the laboratory where it will be centrifuged at 2500 rpm for 15 minutes at 4 degrees centigrade, immediately afterward 500 µl of serum will be aliquoted and stored at minus 75 ° C until later analysis. The general methodology for sandwich ELISA will be used.
Diagnostic Test: Two-dimensional transthoracic echocardiogram — With prior informed consent, a two-dimensional transthoracic echocardiogram will be obtained by an echocardiographer certified by the Mexican Council of Cardiology (CMC) with a Phillips EPIC 7 echocardiography, 2D Arrary 3D Convex (1-6 Mhz) transducer.

SUMMARY:
Background

Calcification of the aortic valve affects more than 26% of adult patients over 65 years of age and is the main indication for valve replacement in the United States of America. Previous evidence shows that aortic valve calcification is an active biological process associated with inflammation. The only actual treatment for severe aortic stenosis is surgical aortic valve replacement (AVR). The materials with which the different types of prostheses are manufactured could induce inflammation per se. Biological prostheses, an incomplete cell removal process and therefore, the presence of residual proteins of animal origin, could induce the immune system's response. In the manufacturing bioprosthesis at the "Ignacio Chávez" National Institute of Cardiology (INC), an evaluation was carried out in the early, and late post-surgical period, it was shown that the inflammatory response after six months is similar to that produced by mechanical prosthesis.

This study's main objective is to evaluate the inflammatory response in patients with post-operated AVR due to biological or mechanical prosthetic valve through different plasma biomarkers in long-term follow-up.

Research question

What is the inflammatory response and calcification in patients who undergo aortic valve replacement for a manufactured prosthesis at the "Ignacio Chávez" National Institute of Cardiology in the long-term follow-up?

Hypothesis

Manufactured bioprostheses at the "Ignacio Chávez" National Institute of Cardiology show a similar or lower inflammatory response to imported bioprostheses or mechanical prostheses associated with less valve dysfunction and more outstanding durability.

DETAILED DESCRIPTION:
Evaluation of the inflammatory response and long-term calcification in post-operated aortic valve replacement patients.

Background

Calcification of the aortic valve affects more than 26% of adult patients over 65 years of age and is the main indication for valve replacement in the United States of America. In Mexico, there is no exact figure for the prevalence and incidence of aortic stenosis. Previous evidence shows that aortic valve calcification is an active biological process, associated with inflammation and increased levels of intracellular adhesion molecule 1 (ICAM-1), pro-inflammatory cytokines such as tumor necrosis factor-alpha (TNF-α), interleukin 6 (IL-6), interleukin 1 (IL-1), interleukin 17 (IL-17), interleukin 18 (IL-18), extracellular matrix proteins (MMP-1), tenascin-C7, osteopontin and bone sialoprotein followed by osteogenic differentiation.

Osteoprotegerin (OPG) / RANK / RANK ligand also plays a regulatory role in bone metabolism; however, in bioprostheses, the role they play in dysfunction does not seem to be clear. They have been found in patients with early coronary atherosclerosis, and a significant increase in endothelial progenitor cells with osteoblasts, osteocalcin (OCN) and phenotype (EPN-OCN) and it has been shown that it is an important prognostic marker in valvular calcification. In the final stage of the disease, expression of TGFβ1 and VAP-1 has been found; both genes are triggers of the calcification process without any association with osteogenic transformation, which is not influenced by statins' use; however, first use alters its expression.

The only actual treatment for severe aortic stenosis is surgical aortic valve replacement (AVR). However, even after the procedure, the inflammatory response persists in almost half of the patients. It has been shown that there is no correlation between age, gender, smoking, ventricular geometry, transvalvular aortic gradient, and the persistence of the inflammatory state after valve replacement. Even more, the materials with which the different types of prostheses are manufactured could induce inflammation per se. Biological prostheses, an incomplete cell removal process and therefore the presence of residual proteins of animal origin, could induce a response of the immune system through the xenoantigen Gal-3-Gal- and its corresponding anti-Gal antibodies that have been associated with valve prosthetic damage. The presence of metallic components such as titanium could act as a trigger for the inflammatory response. As regards the hemodynamic profile of the bioprosthesis, it is unknown whether it is correlated with an inflammatory response. In the manufacturing bioprosthesis at the "Ignacio Chávez" National Institute of Cardiology (INC), an evaluation was carried out in the early, and late post-surgical period, it was shown that the inflammatory response after six months is similar to that produced by mechanical prosthesis.

This study's main objective is to evaluate the inflammatory response in patients with post-operated AVR due to biological or mechanical prosthetic valve through different plasma biomarkers in long-term follow-up.

Problem Statement

The pattern of the inflammatory response and long-term calcification of the prosthetic valve manufactured in the National Institute of Cardiology "Ignacio Chávez" is not known, in the study carried out by Soto López and Cols in which patients undergoing prosthetic valve change were evaluated in a state of early and late post-surgical (6 months) it was observed that there is no difference between biological or mechanical prosthesis. We believe that the inflammatory process associated with the INC bioprosthesis persists over time. However, it could be even less than an imported bioprosthesis or mechanical prosthesis, so it is necessary to evaluate its inflammatory pattern in long-term follow-up.

Justification

Degenerative aortic stenosis is a significant health problem, and its treatment through valve replacement modifies morbidity and mortality. There are currently more than 5000 prostheses implanted in the INC, and the leading cause of dysfunction is calcification. The long-term inflammatory response in INC bioprostheses has not been evaluated to date, identifying, and comparing the inflammatory pattern between these bioprostheses could identify potential therapeutic targets. Demonstrating non-inferiority and a similar or less inflammatory pattern could provide one more reason to start its generalized use in public health institutions in the country.

Research question

What is the inflammatory response and calcification in patients who undergo aortic valve replacement for a manufactured prosthesis at the "Ignacio Chávez" National Institute of Cardiology in the long-term follow-up?

Aims

Primary objectives

• Quantify the long-term inflammatory response of INC bioprostheses implanted in the aortic position.

Secondary objectives

* Compare the long-term inflammatory response of INC bioprostheses implanted in the aortic position to imported bioprostheses and mechanical prostheses.
* The inflammatory response of post-bioprosthesis operated patients will be compared with a control group.

Hypothesis

Null hypothesis

The inflammatory response is more significant in manufactured bioprostheses at the "Ignacio Chávez" National Institute of Cardiology, associated with more significant prosthetic valve dysfunction.

Alternative hypothesis

Manufactured bioprostheses at the "Ignacio Chávez" National Institute of Cardiology show a similar or lower inflammatory response to imported bioprostheses or mechanical prostheses, which is associated with less valve dysfunction and more outstanding durability.

Methodology

Design type

Observational, longitudinal, descriptive ambispective cohort study.

Sample size

The sample size of 56 patients (14 patients per group) was calculated using a test for difference of independent proportions, with a power of 80 %, probability of error of 0.5, based on the RANK concentration from the previous studies.

Statistic analysis.

The normality of continuous variables will be sought with the Shapiro Wilks test. According to the distribution, continuous variables will be expressed as mean ± standard deviation or median and interquartile ranges. The categorical variables will be expressed in number and percentage. Comparisons will be made using the Chi-square test or Fisher's exact test for categorical variables; For dimensional variables, the Student's t-test or Mann-Whitney's U test will be used. The differences will be considered statistically significant when the value of p is less than 0.05.

Schedule of activities.

The preparation of the protocol and review by the ethics committee will be carried out in the months of June to August 2017, the obtaining of the information will take place from August 2017 to February 2018, the obtaining of the inflammatory profile will be carried out in the months of March 2018 to July 2019, the information processing will take place in August and December 2019, the review by the committee will be enhanced in January to July 2020 and the disclosure of results It is carried out during the months of November to December 2020.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age underwent an aortic valve exchange for an INC bioprosthesis, imported bioprosthesis, or mechanical prosthesis.
2. Patients with follow-up two-dimensional transthoracic echocardiography.
3. Patients who agree to take a blood sample for an inflammatory profile.

Exclusion Criteria:

1. Patients in whom more than one cardiac prosthesis was implanted in any valve position.
2. Inflammatory and connective tissue disease (systemic lupus erythematosus, rheumatoid arthritis, antiphospholipid syndrome).
3. Patients undergoing aortic valve replacement due to prosthetic valve dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have had a biological prosthetic valve implanted in aortic position manufactured at the National Institute of Cardiology "Ignacio Chávez" with an anti-calcifying system, imported biological prosthetic aortic valve or mechanical aortic valve from January 1990 to May 2020.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 1990-01-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Quantify the long-term inflammatory response of INC bioprostheses implanted in the aortic position. | An average of 6 years
  Serum measurements of RANK, RANKL, IL-10 (pg/cc), IL-1 (pg/cc), IL-6(pg/cc), ICAM-1 (pg/cc), MMP-9, endothelin-1, osteopontin, osteprogesterin, and TNF-alpha (pg/cc) will be performed.

SECONDARY OUTCOMES:
Compare the long-term inflammatory response of INC bioprostheses implanted in the aortic position to imported bioprostheses and mechanical prostheses. | An average of 6 months
  Serum measurements of RANK, RANKL, IL-10 (pg/cc), IL-1 (pg/cc), IL-6(pg/cc), ICAM-1 (pg/cc), MMP-9, endothelin-1, osteopontin, osteprogesterin, and TNF-alpha (pg/cc) will be performed.
The inflammatory response of post-bioprosthesis operated patients will be compared with a control group. | Through study completion, an average of 6 years
  Serum measurements of RANK, RANKL, IL-10 (pg/cc), IL-1 (pg/cc), IL-6(pg/cc), ICAM-1 (pg/cc), MMP-9, endothelin-1, osteopontin, osteprogesterin, and TNF-alpha (pg/cc) will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elena Soto Lopez, PhD, Principal Investigator — Instituto Nacional de Cardiologia Ignacio Chavez
Locations (1):
- Instituto Nacional Ignacio Chavez, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Lindroos M, Kupari M, Heikkila J, Tilvis R. Prevalence of aortic valve abnormalities in the elderly: an echocardiographic study of a random population sample. J Am Coll Cardiol. 1993 Apr;21(5):1220-5. doi: 10.1016/0735-1097(93)90249-z. PMID 8459080
- [Background] Rajamannan NM. Calcific aortic stenosis: lessons learned from experimental and clinical studies. Arterioscler Thromb Vasc Biol. 2009 Feb;29(2):162-8. doi: 10.1161/ATVBAHA.107.156752. Epub 2008 Nov 20. PMID 19023094
- [Background] Galeone A, Brunetti G, Oranger A, Greco G, Di Benedetto A, Mori G, Colucci S, Zallone A, Paparella D, Grano M. Aortic valvular interstitial cells apoptosis and calcification are mediated by TNF-related apoptosis-inducing ligand. Int J Cardiol. 2013 Nov 15;169(4):296-304. doi: 10.1016/j.ijcard.2013.09.012. Epub 2013 Oct 5. PMID 24148916
- [Background] Kaden JJ, Dempfle CE, Grobholz R, Tran HT, Kilic R, Sarikoc A, Brueckmann M, Vahl C, Hagl S, Haase KK, Borggrefe M. Interleukin-1 beta promotes matrix metalloproteinase expression and cell proliferation in calcific aortic valve stenosis. Atherosclerosis. 2003 Oct;170(2):205-11. doi: 10.1016/s0021-9150(03)00284-3. PMID 14612199
- [Background] Madhur MS, Funt SA, Li L, Vinh A, Chen W, Lob HE, Iwakura Y, Blinder Y, Rahman A, Quyyumi AA, Harrison DG. Role of interleukin 17 in inflammation, atherosclerosis, and vascular function in apolipoprotein e-deficient mice. Arterioscler Thromb Vasc Biol. 2011 Jul;31(7):1565-72. doi: 10.1161/ATVBAHA.111.227629. Epub 2011 Apr 7. PMID 21474820
- [Background] Naito Y, Tsujino T, Wakabayashi K, Matsumoto M, Ohyanagi M, Mitsuno M, Miyamoto Y, Hao H, Hirota S, Okamura H, Masuyama T. Increased interleukin-18 expression in nonrheumatic aortic valve stenosis. Int J Cardiol. 2010 Oct 8;144(2):260-3. doi: 10.1016/j.ijcard.2009.01.022. Epub 2009 Feb 13. PMID 19217172
- [Background] Satta J, Melkko J, Pollanen R, Tuukkanen J, Paakko P, Ohtonen P, Mennander A, Soini Y. Progression of human aortic valve stenosis is associated with tenascin-C expression. J Am Coll Cardiol. 2002 Jan 2;39(1):96-101. doi: 10.1016/s0735-1097(01)01705-3. PMID 11755293
- [Background] Kennedy JH, Henrion D, Wassef M, Shanahan CM, Bloch G, Tedgui A. Osteopontin expression and calcium content in human aortic valves. J Thorac Cardiovasc Surg. 2000 Aug;120(2):427. doi: 10.1067/mtc.2000.106968. No abstract available. PMID 10917976
- [Background] Kaden JJ, Bickelhaupt S, Grobholz R, Haase KK, Sarikoc A, Kilic R, Brueckmann M, Lang S, Zahn I, Vahl C, Hagl S, Dempfle CE, Borggrefe M. Receptor activator of nuclear factor kappaB ligand and osteoprotegerin regulate aortic valve calcification. J Mol Cell Cardiol. 2004 Jan;36(1):57-66. doi: 10.1016/j.yjmcc.2003.09.015. PMID 14734048
- [Background] Caira FC, Stock SR, Gleason TG, McGee EC, Huang J, Bonow RO, Spelsberg TC, McCarthy PM, Rahimtoola SH, Rajamannan NM. Human degenerative valve disease is associated with up-regulation of low-density lipoprotein receptor-related protein 5 receptor-mediated bone formation. J Am Coll Cardiol. 2006 Apr 18;47(8):1707-12. doi: 10.1016/j.jacc.2006.02.040. Epub 2006 Mar 20. PMID 16631011
- [Background] Cao H, Li Q, Li M, Od R, Wu Z, Zhou Q, Cao B, Chen B, Chen Y, Wang D. Osteoprotegerin/RANK/RANKL axis and atrial remodeling in mitral valvular patients with atrial fibrillation. Int J Cardiol. 2013 Jul 1;166(3):702-8. doi: 10.1016/j.ijcard.2011.11.099. Epub 2011 Dec 15. PMID 22178057
- [Background] Gossl M, Modder UI, Atkinson EJ, Lerman A, Khosla S. Osteocalcin expression by circulating endothelial progenitor cells in patients with coronary atherosclerosis. J Am Coll Cardiol. 2008 Oct 14;52(16):1314-25. doi: 10.1016/j.jacc.2008.07.019. PMID 18929243
- [Background] Gossl M, Khosla S, Zhang X, Higano N, Jordan KL, Loeffler D, Enriquez-Sarano M, Lennon RJ, McGregor U, Lerman LO, Lerman A. Role of circulating osteogenic progenitor cells in calcific aortic stenosis. J Am Coll Cardiol. 2012 Nov 6;60(19):1945-53. doi: 10.1016/j.jacc.2012.07.042. Epub 2012 Oct 10. PMID 23062532
- [Background] Anger T, Carson W, Weyand M, Daniel WG, Hoeher M, Garlichs CD. Atherosclerotic inflammation triggers osteogenic bone transformation in calcified and stenotic human aortic valves: still a matter of debate. Exp Mol Pathol. 2009 Feb;86(1):10-7. doi: 10.1016/j.yexmp.2008.11.001. Epub 2008 Nov 19. PMID 19084515
- [Background] Agmon Y, Khandheria BK, Jamil Tajik A, Seward JB, Sicks JD, Fought AJ, O'Fallon WM, Smith TF, Wiebers DO, Meissner I. Inflammation, infection, and aortic valve sclerosis; Insights from the Olmsted County (Minnesota) population. Atherosclerosis. 2004 Jun;174(2):337-42. doi: 10.1016/j.atherosclerosis.2004.01.028. PMID 15136064
- [Background] Anderson JM, Rodriguez A, Chang DT. Foreign body reaction to biomaterials. Semin Immunol. 2008 Apr;20(2):86-100. doi: 10.1016/j.smim.2007.11.004. Epub 2007 Dec 26. PMID 18162407
- [Background] Barone A, Benktander J, Teneberg S, Breimer ME. Characterization of acid and non-acid glycosphingolipids of porcine heart valve cusps as potential immune targets in biological heart valve grafts. Xenotransplantation. 2014 Nov-Dec;21(6):510-22. doi: 10.1111/xen.12123. Epub 2014 Jul 9. PMID 25041314
- [Background] Schanen BC, Karakoti AS, Seal S, Drake DR 3rd, Warren WL, Self WT. Exposure to titanium dioxide nanomaterials provokes inflammation of an in vitro human immune construct. ACS Nano. 2009 Sep 22;3(9):2523-32. doi: 10.1021/nn900403h. PMID 19769402
- [Background] Vesely I. Heart valve tissue engineering. Circ Res. 2005 Oct 14;97(8):743-55. doi: 10.1161/01.RES.0000185326.04010.9f. PMID 16224074
- [Result] Gerber IL, Stewart RA, Hammett CJ, Legget ME, Oxenham H, West TM, French JK, White HD. Effect of aortic valve replacement on c-reactive protein in nonrheumatic aortic stenosis. Am J Cardiol. 2003 Nov 1;92(9):1129-32. doi: 10.1016/j.amjcard.2003.07.012. PMID 14583374
- [Result] Kastellanos SS, Toumpoulis IK, Aggeli C, Zezas S, Chlapoutakis E, Kastellanos S, Stefanadis CI. The role of sex and biochemical markers of inflammation in left ventricular remodelling, before and after surgery, in elderly patients with aortic valve stenosis. Hellenic J Cardiol. 2009 Jan-Feb;50(1):26-36. PMID 19196618
- [Result] Soto ME, Salas JL, Vargas-Barron J, Marquez R, Rodriguez-Hernandez A, Bojalil-Parra R, Perez-Torres I, Guarner-Lans V. Pre- and post-surgical evaluation of the inflammatory response in patients with aortic stenosis treated with different types of prosthesis. BMC Cardiovasc Disord. 2017 Apr 14;17(1):100. doi: 10.1186/s12872-017-0526-1. PMID 28410571
- [Result] Steinmetz M, Skowasch D, Wernert N, Welsch U, Preusse CJ, Welz A, Nickenig G, Bauriedel G. Differential profile of the OPG/RANKL/RANK-system in degenerative aortic native and bioprosthetic valves. J Heart Valve Dis. 2008 Mar;17(2):187-93. PMID 18512489
- [Derived] Saucedo-Orozco H, Vargas-Barron J, Marquez-Velazco R, Farjat-Pasos JI, Martinez-Zavala KS, Jimenez-Rojas V, Criales-Vera SA, Arias-Godinez JA, Fuentevilla-Alvarez G, Guarner-Lans V, Perez-Torres I, Melendez-Ramirez G, Sanchez Perez TE, Soto ME. Bioprosthesis in aortic valve replacement: long-term inflammatory response and functionality. Open Heart. 2022 Aug;9(2):e002065. doi: 10.1136/openhrt-2022-002065. PMID 35926961